CLINICAL TRIAL: NCT03173157
Title: Effect of Targeted Interventions to Improve Value Based Health Care for Inpatient Cardiology Patients: A Choosing Wisely Initiative
Brief Title: Effect of Targeted Interventions to Improve Value Based Health Care for Inpatient Cardiology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Adam Kingeter, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 162135
Record Dates: First submitted 2017-05-25; First posted 2017-06-01 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure; Heart Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Value Feedback Arm (Experimental): A weekly email will be sent to all inpatient, resident-staffed cardiology teams outlining best use practices from AHA/ACC statements on trans-thoracic echoacardiography and data feedback on in-hospital charges, running 13 week average usage and previous week usage of full and limited trans thoracic echocardiograms
  Interventions: Other: Value Feedback Email

INTERVENTIONS:
Other: Value Feedback Email — a biweekly email to three house staff-run cardiology services at VUMC presenting the in-hospital charges and appropriate use of echocardiography. A weekly email will also be sent to the intervention services detailing their team's in-hospital charges for echocardiograms during the preceeding week.

SUMMARY:
The investigators hypothesize that a combined didactic and data feedback program presenting evidence based indications and in-hospital-charges for echocardiograms to inpatient cardiology team members will lead to increased health care value for patients on inpatient cardiology teams.

DETAILED DESCRIPTION:
The cost of healthcare in the United States has risen precipitously over the last forty years. In 2014, healthcare spending surpassed $3 trillion and accounted for 17.5 percent of the national gross domestic product. The Institute of Medicine's report "Best Care at Lower Cost" estimated that 30 percent, or approximately $900 billion in 2014, of healthcare expenditures are wasted. Given this wasted spending, great urgency has been placed on curbing the ever-increasing cost of healthcare while simultaneously improving quality and patient safety. Despite improvements in mortality associated with cardiovascular disease over the last two decades, the cost of cardiovascular care continues to rise and is estimated to be in excess of $186 billion by 2023. A number of studies have been performed evaluating the cost-effectiveness and appropriate use of routine transthoracic echocardiography; nonetheless, there is little evidence that the results of these studies have been translated into clinical practice. In order to close the gap between the literature and clinical practice, we plan to initiate a combined didactic and data feedback program that will present the current literature and in-hospital charges associated with echocardiography to practicing clinicians on inpatient cardiology services. We will measure the effect of our intervention on average per-patient in-hospital charges as well as usage rates and other clinical outcomes.

Research Design and Methods: The investigators will perform a prospective, controlled cohort study period comparing the effect of a combined didactic and data feedback intervention on in-hospital charges, usage rates, and clinical outcomes to providers. The investigator's intervention will consist of a biweekly email to three house staff-run cardiology services at VUMC presenting the in-hospital charges and appropriate use of echocardiography per ACC/AHA guidlines. A weekly email will also be sent to the intervention services detailing their team's in-hospital charges for echocardiograms during the preceding week. Usage and in-hospital charges will be measured using a custom tableau which captures all orders placed in the HeoWiz ordering program and the raw master charges. The investigators will utilize a pre and post intervention design to study primary and secondary outcomes. The primary outcome will be average echocardiography charges per team. The secondary outcomes will be echocardiograms performed per team per month, and number of focused echocardiograms performed per team per month. Quality of care will be assessed by monitoring 30 day readmission rate, and index hospitalization mortality.

ELIGIBILITY:
Inclusion Criteria:

* All residents rotation through inpatient cardiology teams at a large academic medical center

Exclusion Criteria:

* Residents who elect to not recieve feedback email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Average echocardiography charges per inpatient team | 30 days
  Average echocardiography charges per inpatient team per month

SECONDARY OUTCOMES:
Average number of complete transthoracic echocardiograms per inpatient team | 30 days
  Average number of complete transthoracic echocardiograms per inpatient team per month
Average number of focused transthoracic echocardiograms per inpatient team | 30 days
  Average number of focused transthoracic echocardiograms per inpatient team per month

OTHER OUTCOMES:
Readmission rate | 30 day
  Readmission rate for patients admitted to inpatient cardiology teams
Index hospitalization mortality | 30 day
  mortality rate for patients admitted to inpatient cardiology teams

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No